CLINICAL TRIAL: NCT03301298
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Food Effect of SXC-2023 When Administered Orally to Healthy Adult Subjects
Brief Title: Placebo-Controlled Single Dose Study to Evaluate Safety and Pharmacokinetics of SXC-2023 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Promentis Pharmaceuticals, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO-101
Record Dates: First submitted 2017-09-26; First posted 2017-10-04 (Actual); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- SXC-2023, 50 mg (Experimental): Single dose of 50 mg, given orally in capsule form.
  Interventions: Drug: SXC-2023
- SXC-2023, 100 mg (Experimental): Single dose of 100 mg, given orally in capsule form.
  Interventions: Drug: SXC-2023
- SXC-2023, 200 mg (Experimental): Single dose of 200mg, given orally in capsule form.
  Interventions: Drug: SXC-2023
- SXC-2023, 400 mg (Experimental): Single dose of 400mg, given orally in capsule form.
  Interventions: Drug: SXC-2023
- SXC-2023, 800 mg (Experimental): Single dose of 800mg, given orally in capsule form.
  Interventions: Drug: SXC-2023
- SXC-2023, 1600 mg (Experimental): Single dose of 1600 mg, given orally in capsule form.
  Interventions: Drug: SXC-2023
- Placebo oral capsule (Placebo Comparator): Placebo comparator, given once orally in matching capsule form.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: SXC-2023 — Oral capsule
  Arms: SXC-2023, 100 mg; SXC-2023, 1600 mg; SXC-2023, 200 mg; SXC-2023, 400 mg; SXC-2023, 50 mg; SXC-2023, 800 mg
Drug: Placebo oral capsule — Placebo given as oral capsule.
  Arms: Placebo oral capsule

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending oral dose and food effect study conducted at one study center in the United States. Safety and tolerability will be assessed throughout the study and serial blood samples and urine samples will be collected for the safety and pharmacokinetic assessment of SXC-2023.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or females (women of non child bearing potential), 18-55 years of age (inclusive).
2. Medically healthy with no clinically significant screening results.
3. Non-vasectomized male subjects must agree to use birth control or abstain from sexual intercourse during and until 90 days beyond the last dose of study drug/placebo.
4. Continuous non-smoker, at least 3 months prior to first dose and throughout the study.
5. Understands the study procedures in the informed consent form, and be willing and able to comply with the protocol

Exclusion Criteria:

1. Subject is mentally or legally incapacitated.
2. History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subjects by their participation in the study.
3. History or presence of alcoholism or drug abuse within the past 2 years
4. Female subject of childbearing potential.
5. Blood donation or significant blood loss within 56 days prior to first dose.
6. Plasma donation within 7 days prior to first dose.
7. Participation in another clinical trial within 30 days prior to first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tricia Cotter, Study Director — Promentis Pharmaceuticals, Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo comparator, given once orally in matching capsule form.
  Placebo oral capsule: Placebo given as oral capsule.
Period: Unfed Conditions
Arm/Group | SXC-2023, 50 mg | SXC-2023, 100 mg | SXC-2023, 200 mg | SXC-2023, 400 mg | SXC-2023, 800 mg | SXC-2023, 1600 mg | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Fed Conditions
Arm/Group | SXC-2023, 50 mg | SXC-2023, 100 mg | SXC-2023, 200 mg | SXC-2023, 400 mg | SXC-2023, 800 mg | SXC-2023, 1600 mg | Placebo
Started (Only cohort 5 participated in the fed portion of the study, subject 5004 elected to discontinue.) | 0 | 0 | 0 | 0 | 5 | 0 | 2
Completed | 0 | 0 | 0 | 0 | 5 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SXC-2023, 50 mg | SXC-2023, 100 mg | SXC-2023, 200 mg | SXC-2023, 400 mg | SXC-2023, 800 mg | SXC-2023, 1600 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (11.26) | 38 (13.93) | 43.3 (9.35) | 42.8 (14.41) | 38.7 (9.09) | 40 (5.73) | 43.3 (9.43) | 41.3 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 3 | 2 | 3 | 6 | 23
  Male | 3 | 4 | 2 | 3 | 4 | 3 | 6 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 4 | 5 | 5 | 6 | 10 | 37
  Not Hispanic or Latino | 2 | 3 | 2 | 1 | 1 | 0 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3
  White | 5 | 3 | 6 | 6 | 6 | 6 | 11 | 43
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing TEAEs.
Description: Treatment related adverse events as a measure of safety and tolerability of SXC-2023. Measured by patient reporting, assessment of vital signs and laboratory assessments.
Time Frame: 8 days
Measure: Number; unit: participants
Arm/Group | SXC-2023, 50 mg | SXC-2023, 100 mg | SXC-2023, 200 mg | SXC-2023, 400 mg | SXC-2023, 800 mg | SXC-2023, 1600 mg | Placebo Oral Capsule
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
participants | 3 | 0 | 4 | 1 | 2 | 1 | 4

2. Secondary Outcome: Pharmacokinetic Assessments: Cmax
Description: Peak plasma concentration
Time Frame: Samples collected at 0, 1/12, 1/6, 1/4, 1/2, 3/4, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours following dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SXC-2023, 50 mg | SXC-2023, 100 mg | SXC-2023, 200 mg | SXC-2023, 400 mg | SXC-2023, 800 mg | SXC-2023, 1600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 758.2 (157.3) | 2181 (58.3) | 5145 (38.1) | 9005 (60.4) | 25510 (49.5) | 33700 (35)

3. Secondary Outcome: Pharmacokinetics Assessments: Tmax
Description: Time to peak plasma concentration
Time Frame: Samples collected at 0, 1/12, 1/6, 1/4, 1/2, 3/4, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours following dosing.
Population: Subject 1008 who received Treatment A in Cohort 1 did not have any measureable concentration of SXC-2023, NAC, or p-toluic acid and was excluded from the PK population.
Measure: Mean (Full Range); unit: hours
Arm/Group | SXC-2023, 50 mg | SXC-2023, 100 mg | SXC-2023, 200 mg | SXC-2023, 400 mg | SXC-2023, 800 mg | SXC-2023, 1600 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6
hours | 3.111 [3.01 to 4.02] | 3.016 [2.01 to 6] | 4 [2 to 6] | 4 [2 to 4.01] | 2.501 [1.5 to 6] | 3.5 [2 to 4]

4. Secondary Outcome: Pharmacokinetic Assessments: AUC
Description: Area under the plasma concentration-time curve
Time Frame: Samples collected at 0, 1/12, 1/6, 1/4, 1/2, 3/4, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours following dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | SXC-2023, 50 mg | SXC-2023, 100 mg | SXC-2023, 200 mg | SXC-2023, 400 mg | SXC-2023, 800 mg | SXC-2023, 1600 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 3213 (154.1) | 9732 (73.9) | 25180 (43.2) | 57170 (54) | 139500 (28.6) | 239700 (29.8)

5. Secondary Outcome: Pharmacokinetic: Food Effect, AUC
Description: To evaluate the effect of food on the PK of SXC-2023. The log transformed values of total AUC will be analyzed using a linear mixed effect model with formulation, period, sequence, and carryover as fixed effects and subject as a random effect.
Time Frame: Samples collected at 0, 1/12, 1/6, 1/4, 1/2, 3/4, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours following dosing.
Population: Cohort 5 participated in treatment under fasted conditions, followed by treatment under fed conditions. Other Cohorts did not participate.
  Subject 5004 received fasted treatment but discontinued prior to fed treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- SXC-2023, 800 mg Fed: Single dose of 800 mg, given orally in capsule form under fed conditions.
Arm/Group | SXC-2023, 800 mg Fed
Number analyzed (Participants) | 5
ng*hr/mL | 158700 (31.4)

6. Secondary Outcome: Pharmacokinetic: Food Effect, CMax
Description: To evaluate the effect of food on the PK of SXC-2023. The log transformed values of total CMax will be analyzed using a linear mixed effect model with formulation, period, sequence, and carryover as fixed effects and subject as a random effect.
Time Frame: Samples collected at 0, 1/12, 1/6, 1/4, 1/2, 3/4, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours following dosing.
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | SXC-2023, 800 mg Fed
Number analyzed (Participants) | 5
ng/mL | 17160 (26.3)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of subject informed consent through visit followup, approximately 7 days following study drug administration.
Arm/Group | SXC-2023, 50 mg | SXC-2023, 100 mg | SXC-2023, 200 mg | SXC-2023, 400 mg | SXC-2023, 800 mg | SXC-2023, 1600 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 3/6 | 0/6 | 4/6 | 1/6 | 2/6 | 1/6 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SXC-2023, 50 mg (N=6) | SXC-2023, 100 mg (N=6) | SXC-2023, 200 mg (N=6) | SXC-2023, 400 mg (N=6) | SXC-2023, 800 mg (N=6) | SXC-2023, 1600 mg (N=6) | Placebo (N=12)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturation urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT03301298/SAP_000.pdf
  • Study Protocol (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT03301298/Prot_001.pdf